CLINICAL TRIAL: NCT03585101
Title: A Single-arm Evaluation of the Effect of Elbasvir/Grazoprevir on Cardiometabolic Parameters in Patients With Hepatitis C Infection and Underlying Metabolic Disease
Brief Title: A Single-arm Evaluation of the Effect of HCV Treatment on Cardiovascular Disease Risk
Acronym: HEART-C
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding no longer available
Sponsor: University of California, Los Angeles (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kara Chew, Assistant Clinical Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-000650
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus; Endothelial function; Cardiovascular disease risk; Metabolic disease; Inflammation; Insulin resistance
MeSH Terms: conditions — Hepatitis C; Metabolic Diseases; Inflammation; Insulin Resistance | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): Intervention: Elbasvir/grazoprevir
  Interventions: Drug: Elbasvir/grazoprevir

INTERVENTIONS:
Drug: Elbasvir/grazoprevir — Daily fixed-dose combination (FDC) elbasvir (EBR) (50 mg)/grazoprevir (GZR) (100 mg) for 12 weeks
  Other Names: Zepatier, serial number 86336186

SUMMARY:
This study will assess the effect of treatment for hepatitis C virus (HCV) on cardiovascular disease risk. The study will enroll men and women who are infected with HCV and have underlying metabolic disease. All participants will receive a 12-week course of an HCV treatment (elbasvir/grazoprevir). Cardiovascular disease risk will be evaluated at baseline, week 4 on treatment, 12 weeks post-treatment, and 52 weeks post-treatment through noninvasive measurements of endothelial function, insulin resistance, liver fibrosis and steatosis, and circulating blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Presence of HCV infection for at least 12 weeks
* Serum or plasma HCV RNA > lower limit of quantification or detection at any time before or at the time of screening, and the absence of intervening HCV treatment
* Absence of HIV infection
* HCV treatment-naïve OR HCV treatment-experienced with PEG-IFN/RBV only (no prior HCV DAA exposure)
* Genotype 1 or 4 HCV infection. If HCV genotype 1a infection is present, absence of genotype 1a NS5A resistance associated substitutions (RASs) at amino acid positions 28, 30, 31, and 93 must be documented at screening
* Evidence of metabolic disease defined as:

  1. Insulin resistance or impaired glucose tolerance by one of the following:

     * HOMA-IR ≥2.5 at screening
     * Hemoglobin A1c 5.7-6.4% at screening
     * Diabetes mellitus with hemoglobin A1c <7% at screening and never on more than one oral hypoglycemic agent, as well as never requiring insulin

     OR
  2. Metabolic Syndrome, defined as at least 3 of the following:

     * Waist circumference ≥102 cm for men and ≥ 88 cm for women
     * Serum triglyceride level ≥150 mg/dL or on a triglyceride lowering agent
     * Serum high-density lipoprotein (HDL) cholesterol <40 mg/dL in men and <50 mg/dL in women or drug treatment for low HDL cholesterol
     * Blood pressure ≥130/85 mmHg or drug treatment for elevated blood pressure
     * Fasting blood glucose ≥100 mg/dL
* Ability and willingness of subject to provide written informed consent

Exclusion Criteria:

* History of decompensated liver disease (Child Pugh Class B or C)
* Albumin below 3 g/dL
* Platelet count below 75,000
* HBsAg positivity.
* Pregnancy or breastfeeding
* Inability to conform to the following drug interruptions for PAT testing, whether due to safety (determined by the investigator) or willingness: No caffeine or recreational or prescription stimulant use for 24 hours prior; no nicotine for 4 hours prior; no vigorous exercise for 12 hours prior; stopping of beta blockers, short-acting calcium channel blockers (CCBs), nitrates, angiotensin-converting enzyme inhibitors (ACE-Is), angiotensin-receptor blockers (ARBs), and renin-inhibitors for 24 hours prior; and stopping of long acting CCBs 48 hours prior to testing.
* Use of anticoagulant or antiplatelet agents (other than aspirin ≤ 325 mg orally daily) within 1 week prior to study entry or anticipated need for these agents for >7 days during the study follow-up period.
* Use of contraindicated concomitant medications, including OATP1B1/3 inhibitors and strong CYP3A inducers
* Serious illness including acute liver-related disease and malignancy requiring systemic treatment or hospitalization within 12 weeks prior to study entry.
* History of major organ transplantation with an existing functional graft and on immunosuppressive therapy.
* History of known vascular disorder or autoimmune processes including Crohn's disease, ulcerative colitis, severe psoriasis, rheumatoid arthritis, and cryoglobulinemia that may affect vascular studies.
* Decompensated congestive heart failure or acute cardiovascular event (such as stroke, myocardial infarction, arrhythmia, acute peripheral arterial insufficiency) within 6 months prior to study entry
* Use of immune-based therapies or systemic corticosteroids which may affect vascular studies or inflammatory/endothelial biomarkers within 12 weeks prior to study entry
* Advanced renal insufficiency as defined by glomerular filtration rate (GFR) < 30 mL/min/1.73 m2 or treatment by dialysis
* Anticipated inability to comply with research study visits as determined by the investigator
* Poor venous access not allowing screening laboratory collection
* Having any condition that the investigator considers a contraindication to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in reactive hyperemia index (RHI) by peripheral arterial tonometry (PAT) | Baseline to 12 weeks after end of EBR/GZR treatment.

SECONDARY OUTCOMES:
Change in insulin resistance by HOMA-IR | Baseline to 12 weeks after end of treatment
Change in reactive hyperemia index (RHI) by PAT | Baseline to week 4 on treatment
Change in reactive hyperemia index (RHI) by PAT | Baseline to 52 weeks after end of treatment
Change in insulin resistance by HOMA-IR | Baseline to week 4 on treatment
Change in insulin resistance by HOMA-IR | Baseline to 52 weeks after end of treatment
Change in hemoglobin A1c | Baseline to week 4, baseline to 12 weeks after end of treatment, and baseline to 52 weeks after end of treatment
Change in total and LDL cholesterol levels | Baseline to week 4, baseline to 12 weeks after end of treatment, and baseline to 52 weeks after end of treatment
Change in levels of each soluble biomarker (sCD163, sCD14, sICAM-1, PAI-1, sE-selectin, oxidized LDL, Lp-PLA2, and lipoprotein particle quantification) | Baseline to week 4, baseline to 12 weeks after end of treatment, and baseline to 52 weeks after end of treatment
Cross-sectional levels of each soluble biomarker (sCD163, sCD14, sICAM-1, PAI-1, sE-selectin, oxidized LDL, Lp-PLA2, and lipoprotein particle quantification) at each time point for correlation with RHI | Baseline, week 4, post-treatment weeks 12 and 52
Cross-sectional fibrosis score in kPa by transient elastography (TE) for correlation with RHI and soluble biomarkers | Baseline and 12 and 52 weeks after end of treatment
Cross-sectional steatosis score in dB/m by CAP for correlation with RHI and soluble biomarkers at the same time points | Baseline and 12 and 52 weeks after end of treatment
Change in fibrosis score by transient elastography | Baseline to 52 weeks after end of treatment
Change in hepatic steatosis score by CAP | Baseline to 52 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kara W Chew, M.D., M.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA CARE Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No